CLINICAL TRIAL: NCT03995173
Title: Brain Targets for Alcohol Craving in Veterans With mTBI
Brief Title: Pilot rTMS for AUD+mTBI
Acronym: TMS_AUD+mTBI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0949-W; IK2RX000949 (NIH)
Record Dates: First submitted 2019-04-16; First posted 2019-06-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder; Mild Traumatic Brain Injury; Post-traumatic Stress Disorder
Keywords: alcoholism; brain concussion; post-traumatic stress disorder
MeSH Terms: conditions — Alcoholism; Brain Concussion; Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized controlled trial of two parallel groups: active and placebo rTMS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A unblinded member(s) of the research team will be provided with randomization codes from the study biostatistician. A unblended research team member will then provide the PI and rTMS treatment providers with a specific code for the rTMS device. rTMS providers enter the specific rTMS code into the rTMS device and the device is designed to deliver active or placebo rTMS based on this code. The rTMS device is designed to deliver placebo rTMS that looks, sounds and feels like active rTMS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active (Active Comparator): active rTMS
  Interventions: Device: repetitive transcranial magnetic stimulation
- placebo (Placebo Comparator): placebo rTMS
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — rTMS will be delivered with the Magventure MagProX100 with MagOption stimulator and Magpro Cool Coil B65 A/P. The Magpro Cool Coil B65 A/P can be switched to active or placebo (A/P). The Magventure C-B60 coil will be used to deliver single TMS pulses for motor threshold determination.
  Other Names: transcranial magnetic stimulation

SUMMARY:
This is a pilot randomized controlled trial (RCT) for Veteran participants with alcohol use disorder co-occurring with mild traumatic brain injury and/or post-traumatic stress disorder. The treatment intervention is repetitive Transcranial Magnetic Stimulation (rTMS) and the goal is to reduce alcohol craving with this treatment. The study will enroll 20 Veteran participants. Half of these participants will receive real rTMS and half of the participants will receive placebo rTMS. rTMS treatment will be provided over 10 sessions that will occur once every weekday for 2 weeks. Veteran participants will then complete follow-up phone calls to further evaluate alcohol craving and other symptoms.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI), post-traumatic stress disorder (PTSD) and alcohol use disorder (AUD) are high priority disorders for the Department of Veterans Affairs (VA), in part, because these disorders rarely occur in isolation. The co-occurrence compounds brain impairment and negatively impacts symptom presentation and rehabilitation effectiveness. Veterans with co-occurring AUD, mTBI and/or PTSD have few effective treatment options. Thus, treatment development for these Veterans is of great need. The aim of this protocol is to examine safety, feasibility, and the behavioral and neural effects of an repetitive transcranial magnetic stimulation (rTMS) intervention for Veterans with AUD and co-occurring mTBI and/or PTSD. Behavioral and neural effects of rTMS will be examined after the first rTMS session and after the last rTMS session. The investigators hypothesize that the rTMS intervention will be 1) safe, 2) feasible and 3) efficacious. Specifically, the investigators hypothesize that there will be no adverse events related to the rTMS intervention. The investigators hypothesize that all participants enrolled will successfully complete all rTMS sessions. The investigators hypothesize that participants treated with active rTMS, relative to placebo rTMS, will have reduced alcohol craving severity levels. Finally, the investigators hypothesize that participants treated with active rTMS relative to placebo rTMS will have reduced brain activation in response to alcohol cues and improved functional connectivity after the last rTMS session. This is a prospective, pilot, double-blind randomized controlled trial of the intervention rTMS. There will be 2 groups of Veterans with AUD and co-occurring mTBI and/or PTSD those given 1) active rTMS and those given 2) placebo rTMS. Targeted enrollment for this study is 20 Veterans: n=10 active rTMS and n=10 placebo rTMS. Participants will be screened for safety and evaluated on mental health-related behavioral measures. Eligible participants will be randomized to receive active or placebo rTMS. Participants will then complete motor thresholding (MT) to determine rTMS intensity. Participants will then complete 10 sessions of rTMS. These sessions will be completed once daily on week days over two weeks. TMS pulses will be applied to the left DLPFC at 10Hz rate, 4.9 seconds per train, with inter-train interval of 30 seconds, and a total of 20 trains per session. After the 10th rTMS session, participants will complete an MRI which will last approximately 1hour. A sub-sample of participants will complete an MRI immediately after the first rTMS session. Participants will also repeat the mental health behavioral measures after the last rTMS session. Participants will complete follow-up phone interviews to assess for alcohol craving, mTBI symptoms and PTSD symptoms at one day, one week and one month post-rTMS. Completion of this study is an essential first step towards treatment development for Veterans with co-occurring AUD, mTBI and/or PTSD.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Veterans
* Ages 22 through 65
* Meeting AUDIT-C criteria for AUD (4 for men and 3 for women)
* Pass MRI screening using the Center for Translational Imaging (CTI) Safety Form.
* Clinical Institute of Withdrawal Assessment in Alcohol Withdrawal (CIWA-Ar) scores of 10

Exclusion Criteria:

* History of moderate to severe TBI
* Documented and verified history of psychotic spectrum disorders (i.e., schizophrenia, bipolar)
* Receipt of anti-epileptic medications to control active seizures or evidence of documented seizure within past six months
* Receipt of tricyclic anti-depressants, antipsychotic agents, or other drugs that lower the seizure threshold
* Current use of:

  * opiates
  * cocaine
  * amphetamines
  * barbiturates
  * benzodiazepine
  * marijuana/cannabis dependence as determined by the SCID-IV
* Currently prescribed any anti-craving/addiction medications, i.e.:

  * naltrexone
  * varenicline
  * bupropion
  * disulfiram
  * acamprosate
* Meet questionable validity or malingering criteria on the Minnesota Multiphasic Personality Inventory-2-RF (MMPI-2-RF; F: T score 107; F(p): T score 85; TRIN: T score 80; VRIN: T score 80) or the Letter Memory Test (LMT; total score 92%), as determined in IRB#13-077
* Pregnant or nursing
* Have congestive heart failure
* Have cardiac pacemaker or defibrillator, or:

  * cochlear implant
  * nerve stimulator
  * intracranial metal clips
  * implanted medical pump
  * increased intracranial pressure
* History of:

  * surgery on blood vessels in brain and/or valves of the heart
  * brain hemorrhage
  * neurovascular conditions
  * neurodegenerative disorders
  * claustrophobia
  * metal in eye/face
  * shrapnel/bullet remnants in brain
* Actively suicidal as evidenced by plan to harm or recent attempt communicated on the BDI-II or electronic medical record within the past 6 months
* History of mild TBI within the last 3 months

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Penn Alcohol Craving Scale Change | baseline, immediately after last/10th rTMS session, and 1 day, 1 week, and 1 month follow-up
  5-item self-report measure of alcohol craving and each item is scored on a scale of 0 to 6. The minimum total score is 0 and the maximum is 30, indicating less to more severe alcohol craving, respectively.
Total Adverse Event Frequency | immediately after last/10th rTMS session - up to 2 weeks
  An adverse event log will be kept for each participant and each rTMS treatment session. After each treatment these events will be recorded and the total frequency of events will be used as the outcome after all 10 rTMS sessions over the course of the 2 week treatment have been completed.
Total rTMS Sessions Completed | after the 10th and last rTMS treatment session - up to 2 weeks
  Total number of rTMS treatment sessions completed out of 10 sessions. After all 10 rTMS sessions over the course of the 2 week treatment this cumulative total number of sessions complete can be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Herrold, PhD BA, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT03995173/ICF_000.pdf